CLINICAL TRIAL: NCT06955845
Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) Therapy Versus Selective Serotonin Reuptake Inhibitors (SSRIs) in the Treatment of Post-Traumatic Stress Disorder: A Randomized Controlled Trial
Brief Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) Therapy Versus Selective Serotonin Reuptake Inhibitors (SSRIs) in the Treatment of Post-Traumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asad Ullah Jan (Other Government)
Collaborators: CMH Nowshera (Unknown)
Responsible Party: Sponsor-Investigator, Asad Ullah Jan, Consultant Psychiatrist, Combined Military Hospital Nowshera
Organization: Combined Military Hospital Nowshera (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMHNSR-REF-14
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: PTSD; PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; EMDR; SSRIs; Trauma; Mental Health; Randomized controlled trial; Post-traumatic stress disorder; Eye Movement Desensitization and Reprocessing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Wounds and Injuries; Psychological Well-Being | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR Therapy (Experimental): Participants will receive Eye Movement Desensitization and Reprocessing (EMDR) therapy over six weeks.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing Therapy
- Selective Serotonin Reuptake Inhibitors (SSRIs)Treatment (Active Comparator): Participants will receive selective serotonin reuptake inhibitors (SSRIs) such as Sertraline over six weeks.
  Interventions: Drug: Selective serotonin reuptake inhibitors

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing Therapy — Patients in this arm will receive weekly EMDR sessions for 6 weeks
  Other Names: EMDR Therapy
  Arms: EMDR Therapy
Drug: Selective serotonin reuptake inhibitors — The patients will receive an SSRI medication daily for 6 weeks. The dose will be titrated by the clinician.
  Arms: Selective Serotonin Reuptake Inhibitors (SSRIs)Treatment

SUMMARY:
This randomized controlled trial aims to compare the efficacy of Eye Movement Desensitization and Reprocessing (EMDR) therapy versus Selective Serotonin Reuptake Inhibitors (SSRIs) in the treatment of Post-Traumatic Stress Disorder (PTSD). Adult patients diagnosed with PTSD will be randomly assigned to receive either EMDR therapy or SSRIs for a period of six weeks. The primary outcome is the rate of remission as measured by validated PTSD symptom severity scales at Week 6. Secondary outcomes include changes in functional impairment and patient-reported quality of life. The study seeks to determine whether EMDR therapy is a non-pharmacological alternative to SSRIs for achieving symptom remission in PTSD.

ELIGIBILITY:
Inclusion Criteria:

Age 18-60 years

Clinical diagnosis of Post-Traumatic Stress Disorder (PTSD)

Duration of illness ≥ 6 months

Able to provide informed consent

Exclusion Criteria:

Current substance abuse or dependence

History of psychotic disorder or bipolar disorder

Active suicidal ideation

Concurrent psychotherapy or psychiatric medication (except study-assigned SSRI)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate at Week 6 | 6 weeks
  Each group's proportion of participants achieving remission from PTSD is defined as having a score below 22 on the PTSD Checklist for DSM-5 (PCL-5; range 0-80, where higher scores indicate worse PTSD symptoms), a validated PTSD scale.

SECONDARY OUTCOMES:
Change in functional impairment score | 6 weeks
  Change from baseline to 6 weeks in functional impairment as measured by the World Health Organization Quality of Life-BREF (WHOQOL-BREF; range 26-130, higher scores = better quality of life), a validated quality of life scale.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Ullah Jan, MBBS,FCPS, Principal Investigator — CMH Nowshera
Locations (2):
- Pakistan (2):
  - Combined Military Hospital, Nowshera, KPK
  - Department of Psychiatry, Combined Military Hospital Nowshera, Nowshera, Kpk

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD at this time.